CLINICAL TRIAL: NCT05912257
Title: Preserving Physical Function in Older Adults With Cancer: Impact of an Optimizing Nutrition Intervention Applied Before and After Surgery
Acronym: NOSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F3981-R
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Surgery; Perioperative Nutrition; Older Adults
MeSH Terms: conditions — Neoplasms | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NOSH (Experimental): Multi-Targeted NOSH + Exercise (NOSH Regimen) Arm
  Interventions: Behavioral: Structured perioperative nutrition and exercise
- Typical Regimen (Active Comparator): Typical Regimen Arm
  Interventions: Behavioral: Nutrition and Exercise Counseling

INTERVENTIONS:
Behavioral: Structured perioperative nutrition and exercise — Nutrition counseling by a RD and prescribed a eucaloric diet with protein intake of 1.5 g/kg/d and at least 30 g high quality protein per meal. They will be provided 30 grams of high quality protein twice a day, Hydroxymethylbutyrate, and vitamin D3 and multi-vitamin. Participants will attend nutrition and exercise group classes 6-8 weeks. Following following discharge home, participants will be instructed to resume group classes and protein, HMB, vitamin-D and MVS regimen, and exercise classes will resume when cleared by surgical team.
  Arms: NOSH
Behavioral: Nutrition and Exercise Counseling — nutrition counseling by study Registered Dietitian (RD) and prescribed a eucaloric diet with protein intake of 1.0 g/kg/d and a one a day multivitamin/multimineral supplement. They will be counseled on exercising three times per week and given access to exercise videos. Following following discharge home, participants will be instructed to resume protein recommendations and MVS, and exercise recommendations will resume when cleared by surgical team.
  Arms: Typical Regimen

SUMMARY:
In this pragmatic clinical trial, the investigators will study older Veterans approaching surgery for gastrointestinal or genitourinary cancer who are at high risk for a marked decline in their physical function. The investigators will test a multi-targeted nutrition regimen high in protein and other key nutrients and including resistance exercise, administered 8 weeks prior to surgery and for 24 weeks after discharge from surgery, with the goal of protecting physical function and improving physiologic, metabolic, and patient-centered outcomes. The findings of this study will promote a better intervention to compensate for the high nutritional demands of cancer and its treatment and lead to stronger, more rapid physical recoveries and better quality of life for older adults with moderate to advanced cancer-a group that has rarely been included in long-term nutrition studies. In addition to providing direct benefits to Veterans, the study may also benefit the VA by decreasing demands on the health care system via hastening the recovery of physical function.

DETAILED DESCRIPTION:
The overall objective of this study is to administer the nutrition optimization of senior health (NOSH) intervention in biphasic intervals and compare it to a typically recommended nutrition regimen (Typical Regimen) for (1) physical function, (2) physiologic and metabolic outcomes; and (3) Veteran-centered outcomes. The central hypothesis is that NOSH will improve physical function. The investigators also predict improvements in physiologic, metabolic and Veteran-centered outcomes. The investigators seek an optimal intervention to alleviate symptom burden and improve function, health, and QoL for older cancer survivors, and the long-term goal is to confirm and implement this intervention. The primary aim is to evaluate the efficacy of a multi-targeted NOSH intervention on physical function. Based on preliminary data, the investigators' working hypothesis is that the NOSH intervention will result in improved physical function before surgery and after surgery relative to the (Typical Regimen).

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Veterans
* Stage I, II, III cancer of the bladder, colon, kidney, liver, pancreas, stomach or rectum
* Surgery 6 weeks from consent
* Age > 60 years
* Age-normal renal function
* English speaking
* Able to record dietary intake or has a proxy who can record dietary intake
* Willing and able to be randomized to either intervention group

Exclusion Criteria:

* Stage IV cancer diagnosis
* Glomerular filtration rates (GFR) less than 45 mL/min
* Neurological conditions causing functional impairments, including Parkinson's disease, multiple sclerosis, and permanent disability due to stroke
* Class III-IV congestive heart failure
* Refractory cachexia - medical condition that affects ability to increase muscle mass (e.g., cachexia) defined as 10% weight loss in 10 months, 5% weight loss in 6 months or 2% weight loss over any period plus body mass index 20 kg/m2 AND Life expectancy 9 months
* Active treatment for another cancer site
* Body weight >450 lbs
* Uncontrolled diabetes (HbA1c 9%)
* Recent diagnosis of thyroid disease or untreated thyroid disease
* Inability to complete physical function assessment
* Severe dietary restrictions
* On chemotherapy drug Sorafenib

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Change | baseline, within 24 hours before surgery, 30-days post-op, 12-weeks following post-op visit, 24 weeks following post-op visit
  Distance walked in 6 minute.

SECONDARY OUTCOMES:
Health-related QoL (QLQ-C30) | baseline, within 24 hours before surgery, 30-days post-op, 12-weeks following post-op visit, 24 weeks following post-op visit
  QLQ-C30 is a patient reported outcome measure designed to assess the functional health (physical, role, emotional, social, cognitive), symptom burden (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, dyspnea), and health-related quality of life of adults with cancer. Raw scores are transformed to a 0-100 scale, with a higher score representing better functioning/quality of life and greater symptom burden.
Patient Generated-Subjective Global Assessment (PG-SGA) | baseline, within 24 hours before surgery, 30-days post-op, 12-weeks following post-op visit, 24 weeks following post-op visit
  PG-SGA is a hands-on assessment of weight, muscle and fat mass, food intake, and nutrition impact symptoms117 using a global rating nutritional diagnosis (A=well nourished, B = moderate/suspected malnutrition, or C=severely malnourished) and a continuous numerical score (1 to 30 - with higher scores representing greater nutritional risk) for intervention triage. The continuous numerical score allows for comparison of changes in nutritional status over short duration of time.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn N. Starr, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No